CLINICAL TRIAL: NCT00061607
Title: SMN Levels in Peripheral Blood Samples of SMA Patients and the Effects of Pharmacological Compounds In Vitro
Brief Title: Measuring Levels of SMN in Blood Samples of SMA Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030203; 03-N-0203
Record Dates: First submitted 2003-05-29; First posted 2003-05-30 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Motor Neuron Disease; Neuromuscular Disease; Histone Deacytelase Inhibitors; Spinal Muscular Atrophy; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal; Motor Neuron Disease; Neuromuscular Diseases

SUMMARY:
Spinal muscular atrophy (SMA) is a disorder that affects the motor neurons. SMA is caused by a mutation in a part of the DNA called the survival motor neuron (SMN1) gene, which normally produces a protein called SMN. Because of their gene mutation, people with SMA make less SMN protein, which results in the loss of motor neurons. SMA symptoms may be improved by increasing the levels of SMN protein. The purpose of this study is to determine whether a drug called a histone deacetylase inhibitor can increase SMN levels.

After undergoing a general medical and neurological evaluation, study participants will donate a blood sample. Researchers will use this sample to measure SMN levels. They will also isolate cells from the blood and treat the cells with various drugs that may increase SMN levels.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a currently untreatable, autosomal recessive motor neuron disease that is caused by deficiency of full-length survival motor neuron (SMN) protein. One promising therapeutic approach to SMA is to pharmacologically increase full-length SMN protein levels. Several compounds have been shown to increase SMN levels in immortalized cell lines derived from SMA patients. The objective of this study is to determine baseline SMN levels in primary peripheral blood cells of SMA patients and heterozygous carriers compared to unaffected controls and to investigate the effects in vitro of pharmacological compounds that are expected to increase SMN levels. It is anticipated that these studies will provide further evidence to support the use of one or more of these compounds in a clinical trial for SMA patients. The study population will include patients with genetically proven type I, II, or III SMA and their family members. Blood samples from anonymous, unaffected control patients will be obtained through the department of transfusion medicine (99-CC-0168). This is an investigative study that involves blood drawing only. No new therapy will be provided except the standard of care.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of SMA with genetically proven mutations in the SMN1 gene or unaffected family members (age greater than or equal to 2 years).

No exposure to valproic acid or any other HDAC inhibitors for a period of at least 2 weeks.

Written, informed consent (and assent, if applicable).

EXCLUSION CRITERIA:

History of valproic acid or other HDAC inhibitor use within the past14 days.

History of bleeding disorder, which would make a blood draw unsafe.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-05-19; Study Completion 2017-04-04

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Crawford TO, Pardo CA. The neurobiology of childhood spinal muscular atrophy. Neurobiol Dis. 1996 Apr;3(2):97-110. doi: 10.1006/nbdi.1996.0010. No abstract available. PMID 9173917
- [Background] Pearn J. Incidence, prevalence, and gene frequency studies of chronic childhood spinal muscular atrophy. J Med Genet. 1978 Dec;15(6):409-13. doi: 10.1136/jmg.15.6.409. PMID 745211
- [Background] Nicole S, Diaz CC, Frugier T, Melki J. Spinal muscular atrophy: recent advances and future prospects. Muscle Nerve. 2002 Jul;26(1):4-13. doi: 10.1002/mus.10110. PMID 12115944